CLINICAL TRIAL: NCT00187343
Title: A Phase III Study of Adjuvant Radiation Therapy in Early Breast Cancer Comparing the Use of Breast Intensity Modulated Radiation Therapy (IMRT) to Conventional Wedge Technique
Brief Title: A Clinical Trial to Reduce Skin Burn Induced by Breast Radiotherapy Using Intensity Modulated Radiation Therapy (IMRT)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: British Columbia Cancer Agency (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BreastIMRT
Record Dates: First submitted 2005-09-12; First posted 2005-09-16 (Estimated); Last update posted 2008-09-08 (Estimated); Status verified 2005-09

CONDITIONS: Breast Neoplasms
Keywords: Radiotherapy; IMRT
MeSH Terms: conditions — Breast Neoplasms

INTERVENTIONS:
Device: Breast IMRT

SUMMARY:
The purpose of this study is to determine whether the use of a 3D missing tissue compensation radiation technique during a standard adjuvant breast radiotherapy delivering a dose of 50Gy in 25 treatments could reduce significantly the occurence rate and the degree of acute skin reaction compared to a standard wedged irradiation technique.

DETAILED DESCRIPTION:
1. Description of the Problem:

   The majority of breast cancer patients are treated with breast-conserving surgery followed by radiotherapy, giving loco-regional control rates similar to mastectomy. Currently, the "standard" breast radiotherapy technique includes treatment of the entire breast with a tangential opposed pair of photon beams. The standard technique leads to significant acute skin toxicity, ranging from breast erythema to moist desquamation, in approximately 40% of patients. This toxicity may lead to interruptions in treatment delivery; may increase the risk of developing late skin toxicity including telangiectasia, skin fibrosis and chronic breast pain; and may also be associated with a significant decrease in health-related quality of life (HRQOL). Published data from dosimetric studies suggest that dose variations in excess of 10% within the breast may be the most important predictor of acute radiation-induced skin toxicity (RR = 9.7), and that dose toxicity occurs more frequently in the inframamary fold. A study performed at TSRCC shows that intensity modulated radiotherapy (IMRT) allows for significant improvements in dose homogeneity within the breast compared to standard breast radiotherapy techniques. Furthermore, the hot spot over 10% seen in the inframamary fold for patient with large breast volume is removed.
2. Objectives:

   * To determine if the occurence of acute skin toxicity in women receiving adjuvant breast radiation with IMRT is less frequent compared to women treated with conventional technique.
   * To determine if the HRQOL scores, and specifically breast module subscale scores, in women receiving adjuvant breast radiation with IMRT is better than HRQOL scores in women receiving conventional technique.
   * To perform a comparison of costs in the delivery of breast radiotherapy using IMRT to conventional technique.
   * To determine if an increased acute skin toxicity translates into an increased late skin toxicity.
3. Hypothesis:

We hypothesize that women receiving adjuvant breast radiation with IMRT will have significantly less acute skin toxicity and improved HRQOL compared to women treated with conventional techniques. We also hypothesize that there would not be increased cost related to IMRT compared to conventional technique.

Research plan: A Phase III randomised controled trial is planned, with blocked stratification on breast size and boost delivery. Eligible women include those who have been referred to TSRCC following breast-conserving surgery. They will be randomized to receive either a conventional technique treatment, either breast IMRT. Acute skin toxicity will be assessed weekly during radiotherapy and up to one month following completion of radiotherapy using the previously validated RTOG acute skin toxicity scale. The occurence, duration and intensity of acute skin toxicity will be compared. HRQOL will be assessed during and after irradiation, using validated EORTC instruments (EORTC QLQ-C30 and QLQ-BR23). 340 patients will be accrued in order to detect a 15% reduction in the ocurence of acute skin toxicity with IMRT using an a=0.05, b=0.80.

ELIGIBILITY:
Inclusion Criteria:

* A confirmed histological diagnosis of breast carcinoma or DCIS;
* Treated by breast conserving surgery;
* Adjuvant radiation to the breast only (less than 3 positive lymph nodes);
* Having a ECOG performance status of 0 or 1.
* Having signed an informed consent.

Exclusion Criteria:

* Patients treated by mastectomy;
* Bilateral breast cancer;
* Having an unhealed surgical scar (skin not closed and/or infection);
* Having had prior radiation to the same breast;
* Having active connective tissue disorder;
* Patient being pregnant.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 340
Dates: Start 2003-09; Study Completion 2005-06

PRIMARY OUTCOMES:
Maximum skin toxicity measured weekly during the tratment and bi-weekly up to one month after the end of the treatment and complete resolution of skin reaction using the NCI common toxicity criteria version 3.0 scale

SECONDARY OUTCOMES:
Breast localisation of maximum acute skin toxicity;
Time of onset of acute skin toxicity;
Pain assessment;
Duration of symptoms;
Factors associated with acute skin reactions;
HRQOL;
Drug prescription for skin care.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Philippe PIGNOL, MD, PhD, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (2):
- Canada (2):
  - BC Cancer Agency-Vancouver Island Centre, Victoria, British Columbia
  - Sunnybrook and Women's College Health Sciences Centre, Toronto, Ontario

REFERENCES:
- [Background] Mihai A, Rakovitch E, Sixel K, Woo T, Cardoso M, Bell C, Ruschin M, Pignol JP. Inverse vs. forward breast IMRT planning. Med Dosim. 2005 Fall;30(3):149-54. doi: 10.1016/j.meddos.2005.03.004. PMID 16112466
- See also: Facility information — http://www.sunnybrook.ca/